CLINICAL TRIAL: NCT04565704
Title: Optical Imaging of Gastrointestinal Biopsy Samples and Their Correlation With Histology
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator - MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015P000328
Record Dates: First submitted 2020-08-11; First posted 2020-09-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Gastrointestinal Disease; Gastrointestinal Dysfunction
Keywords: OCT; Optical Coherence Tomography; Biopsy; GI disease; Endoscopy screening; Endoscopic Screening
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Development of novel optical imaging technologies (Experimental): Consented participants will allow their endoscopist to collect 3 additional biopsies from the participants. These biopsies will be used to develop our imaging techniques at our lab. We will use the standard of care histology images from the endoscopy procedure as a control comparison.
  Interventions: Device: Biopsy imaged by Optical imaging device.

INTERVENTIONS:
Device: Biopsy imaged by Optical imaging device.

SUMMARY:
To develop novel optical imaging technologies for use as a non-destructive and minimally invasive tool for detection and diagnosis of various diseases that affect the gastrointestinal system.

DETAILED DESCRIPTION:
The investigators have previously developed optical imaging systems that have been able to provide highly detailed images of tissue structures in multiple application areas including Cardiology, Gastroenterology, and Pulmonology. They are looking to continue the advancement of these various technologies under development.

The population will include participants who are undergoing elective esophagogastroduodenoscopy with biopsy, colonoscopy with biopsy, and/or endo-mucosal resection.The endoscopist will take no more than 3 biopsies in addition to the standard of care biopsies.

The study will be optical imaging of the ex vivo GI specimens that are being collected. Specimens will be collected for research purposes only. Offline analysis of the samples will be performed, and optical imaging findings will be correlated with the pathology findings. This will require review of the medical record to link the findings of the imaging with the pertinent medical information. Samples will be de-identified and participants will be assigned a unique number. The tissues will be placed in marked containers labeled "for research purposes only". The samples collected will be brought to the Tearney Research Laboratory for imaging and processing. The Optical imaging of the tissue samples will not affect the standard of care procedure.

ELIGIBILITY:
Inclusion Criteria:

• Scheduled for an elective esophagoduodenoscopy and/or colonoscopy

Exclusion Criteria:

• According to standard of care at MGH endoscopy department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-03-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Feasibility based on image quality and presence of microscopic features | Imaging data is collected during the procedure, and analyzed within 1 year of collection.
  The feasibility will be determined by at least one of the following parameters: 1) assessing image adequacy (resolution, contrast, etc.) qualitatively, 2) confirming that microscopic features observed in the images are also seen by correlative histopathology, 3) ability to develop preliminary criteria or algorithms based on image-histopathology matches.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No